CLINICAL TRIAL: NCT03938662
Title: Randomised Controlled Trial Assessing the Effect of S-adenosylmethionine Plus Choline in Treatment of Patients With Alcoholic Liver Disease
Brief Title: S-adenosylmethionine Plus Choline in Treatment of Patients With Alcoholic Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Clinic Dr Dragisa Misovic-Dedinje (Other)
Responsible Party: Principal Investigator, Nikola Panic, Principal investigator, University Clinic Dr Dragisa Misovic-Dedinje
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCDragisaMisovic
Record Dates: First submitted 2019-04-30; First posted 2019-05-06 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Alcoholic Liver Diseases
Keywords: alcoholic liver diseases; S-Adenosyl methionine; choline
MeSH Terms: conditions — Liver Diseases, Alcoholic | interventions — Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-Adenosyl methionine and choline (Experimental): Patients in will be administered with formulation of 100 mg of S-Adenosyl methionine and 82.5 mg of choline, once daily for 24 weeks.
  Interventions: Dietary Supplement: formulation containing S-Adenosyl methionine and choline
- Placebo (Placebo Comparator): Patients in will be administered with placebo once daily for 24 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: formulation containing S-Adenosyl methionine and choline — Patients will be administered with formulation containing S-Adenosyl methionine and choline once daily for the period of 24 weeks.
  Arms: S-Adenosyl methionine and choline
Dietary Supplement: Placebo — Placebo of same appearance, colour and taste,
  Arms: Placebo

SUMMARY:
The study will assess the effect of treatment with formulation containing S-Adenosyl methionine and choline, on patients with alcoholic liver disease.

Half of the patients included will receive named formulation once daily for 24 weeks while other half will receive placebo.

DETAILED DESCRIPTION:
Choline and S-Adenosyl methionine are nutrients both showing hepatoprotective effects.

Choline helps liver metabolise glucose and lipids and repair cell membrane. S-Adenosyl methionine is essential for the synthesis of glutathione, a main cellular antioxidant showing its protective effect against free radicals, among others in liver tissue. Furthermore S-Adenosyl methionine is involved in regulation of hepatocyte growth, differentiation, and death. It also enables endogenous production of small amount of choline. Although human organism has capacity for production of small amount of S-Adenosyl methionine, damaged liver can not produce it or produce it insufficient amounts.

Having this in mind it can be hypothesised that administration of choline and S-Adenosyl methionine can be beneficial in patients with alcoholic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* alcoholic liver disease

Exclusion Criteria:

* hepatitis B
* hepatitis C
* autoimmune hepatitis
* hemochromatosis
* Wilson's disease
* hepatocellular carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Alanine aminotransferase (ALT) | 24 weeks
  Alanine aminotransferase will be measured at the enrolment and after 24 weeks of treatment.

SECONDARY OUTCOMES:
Aspartate aminotransferase (AST) | 24 weeks
  Aspartate aminotransferase will be measured at the enrolment and after 24 weeks of treatment.
Gamma-glutamyl transferase (GGT) | 24 weeks
  Gamma-glutamyl transferase will be measured at the enrolment and after 24 weeks of treatment.
Alkaline phosphatase (ALP) | 24 weeks
  Alkaline phosphatase will be measured at the enrolment and after 24 weeks of treatment.
Serum bilirubin | 24 weeks
  Bilirubin levels will be measured at the enrolment and after 24 weeks of treatment.

OTHER OUTCOMES:
Serum proteins | 24 week
  Serum proteins will be measured at the enrolment and after 24 weeks of treatment.
Serum albumins | 24 week
  Serum albumins will be measured at the enrolment and after 24 weeks of treatment.
Serum cholesterol | 24 week
  Serum cholesterol will be measured at the enrolment and after 24 weeks of treatment.
Serum triglycerides | 24 week
  Serum triglycerides will be measured at the enrolment and after 24 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic Dr Dragisa Misovic-Dedinje, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No